CLINICAL TRIAL: NCT00389402
Title: A Randomised, Controlled, Open-Label, 48-Week, Study To Asses Differences in Changes In Plasma Lipid Profile Between Patients On Saquinavir/Ritonavir Or Atazanavir/Ritonavir In Combination With Tenofovir Disoproxil Fumarate And Emtricitabine As A First-line Regimen.
Brief Title: BASIC: Boosted Atazanavir or Saquinavir Induced Lipid Changes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Antiviral Therapy Evaluation Center (Other)
Collaborators: Hoffmann-La Roche (Industry); Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-IAT-0110; Eudract number: 2006-000666-37
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infections
Keywords: lipids; lipodystrophy; fat distribution; hiv-1; antiretroviral therapy; Treatment Naive
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Acquired Immunodeficiency Syndrome | interventions — Saquinavir; Ritonavir; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: saquinavir/ritonavir
Drug: atazanavir/ritonavir

SUMMARY:
The purpose of this study is to assess differences in changes in plasma lipids between patients on saquinavir/ritonavir or atazanavir/ritonavir in combination with tenofovir disoproxil fumarate and emtricitabine as a first-line regimen in patients previously naive for antiretroviral therapy. This study is an extension from the SSAR 2004/0002 which randomised patients over the same treatment arms.

DETAILED DESCRIPTION:
The main objective of the study is to measure changes in blood lipids during 48 weeks of treatment with saquinavir (SQV) / ritonavir (RTV) or atazanavir (ATV) / RTV, in combination with tenofovir (TDF) / emtricitabine (FTC). All of these medications are commonly used for the treatment of HIV-1 infection. When the initial anti-HIV therapy is selected, several important issues are considered such as the effectiveness, the possible long- and/or short-term side effects, the frequency of medication intake and the amount of pills that needs to be taken.

There is currently some concern about the long-term metabolic side effects of existing treatment regimens. Metabolic disorders, such as elevated blood lipids (including cholesterol) and a decreased sensitivity for insulin, which increases the chance of diabetes, pose an increased risk of cardiovascular disease. A large cohort study (the D:A:D study), executed worldwide, including in Dutch hospitals, has actually shown that the use of HIV combination therapy coincides with an increased risk of developing cardiovascular disease. A certain category of HIV inhibitors, the protease inhibitors, are particularly associated with elevated blood lipids. Results from the afore-mentioned worldwide study have recently indicated that in particular the use of protease inhibitors increases the risk of cardiovascular disease, which can to an important extent be explained by a change in the blood lipids caused by these medications. There are however some protease inhibitors, such as the recently developed drug atazanavir (ATV) and the protease inhibitor saquinavir (SQV) that has already been available for several years, which show no to only a little effect on blood lipids. SQV had the disadvantage of having to be dosed twice-daily, with many capsules (10-12 in total per day). Now that a new SQV tablet has been developed, the number of capsules to be taken per day has decreased dramatically (to only 4 in total per day) and moreover it has become possible in actual practice to take these capsules once per day. It is advisable, for both SQV and ATV, to combine the medication with one capsule of ritonavir (RTV), another protease inhibitor. This ensures that a reliable and effective level of SQV or ATV will be reached in the blood. RTV is associated with elevated blood lipids, but this effect is very limited in the low dosage that is used in combination with ATV or SQV. And as both SQV and ATV are combined with an equal amount of RTV, it is expected that their favorable effect on the blood lipids will be the same. For the same reason, the risk of cardiovascular disease is expected to be equally limited with the use of either of these two regimens.

In addition to long-term effects on the blood lipids, which poses a risk of cardiovascular disease, a disturbed fat distribution (lipodystrophy) is another frequently occurring complication in the treatment of HIV-1 infection. This disturbed fat distribution is associated with subcutaneous fat loss in some body parts (particularly the face, arms and legs, and buttocks) and with fat accumulation in other body parts (such as the abdomen, the back of the neck and female breasts). Subcutaneous fat loss is mainly associated with thymidine-containing nucleoside analogues like zidovudine (AZT) and stavudine (d4T). Previous studies in patients receiving antiretroviral treatment for the first time have shown that a combination of TDF / lamivudine (3TC) (the latter drug closely resembles FTC) does not lead to loss of subcutaneous fat (lipoatrophy), as opposed to the combination d4T / 3TC or AZT / 3TC. The cause of fat accumulation is however less clear, but often coincides with changes in blood lipids. The chance of the occurrence of fat accumulation could thus depend on the extent to which an HIV combination therapy coincides with an elevation of blood lipids.

As it is now becoming clear that there are initial therapies involving less risk of long-term side effects, it is important to develop therapy schedules that are safe with regard to these aspects. According to what has been described before, a combination of either ATV / RTV or SQV / RTV, administered together with TDF and FTC to prevent fat loss, would be a good initial regimen, as these combinations have little to no effect on the blood lipids and may therefore decrease the chance of fat accumulation. A big advantage of the use of combination therapy with protease inhibitors in combination with a low dose of RTV is that it largely diminishes the chance of the development of resistance to HIV protease inhibitors, even if the virus becomes detectable in the blood again after initial suppression - as opposed to the most commonly used alternative initial therapy in which non-nucleoside reverse transcriptase inhibitors are used instead of protease inhibitors. With the use of these drugs, the risk of resistance is much greater. It is therefore essential to better examine these protease-inhibitor-containing regimens, which are expected to have the advantage of producing a minimal effect on the lipid and sugar metabolism as well as a limited chance of resistance development.

In the BASIC study we want to show that SQV / RTV is comparable to ATV / RTV with regard to the effect on blood lipids. We will also look in detail at the effects on fat loss and fat accumulation, as well as on sugar metabolism and insulin sensitivity, in the hope that only very limited changes in these areas will be demonstrated.

One study in which patients were given their first antiretroviral treatment demonstrated a slight decrease in bone density (a form of bone loss) in the first year of treatment with TDF and FTC (which closely resembles 3TC). This did however not cause any clinical problems. It was very reassuring to see that a complete recovery of the bone density was again seen after this first year. Nevertheless we want to collect more data about the possible effects on the bone metabolism and for this reason we will perform two bone density assessments during this study. Finally, there are indications that the renal function in patients who are treated with TDF may become slightly disturbed. It is as yet not clear which method can most accurately estimate and detect these slight changes in renal function. For this reason, we plan to compare a number of different methods to estimate renal function as part of this study. For this purpose a number of additional relevant measurements will be obtained using the blood samples which are already being collected as part of the study anyway.

The main purpose of the study is to measure changes in the blood lipids and to compare these between patients who start with either an SQV / RTV-containing regimen or an ATV / RTV-containing regimen. In addition, the changes in fat distribution, sugar metabolism and insulin sensitivity will be compared between these groups. Possible changes in bone density and renal function will also be examined. Furthermore, the virologic effectiveness and overall safety of the two treatments will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Providing written informed consent
* HIV-1 infected patients.
* At least 18 years of age.
* Males or non-pregnant, non-lactating females. Women of childbearing age must have a negative urine pregnancy test at screening. All female participants must be encouraged to utilise adequate contraception for the month preceding entry and for the duration of the study.
* Anti-retroviral treatment naive.
* Indication for antiretroviral therapy according to current treatment guidelines.

Exclusion Criteria:

* CD4 count > 350 cells/mm3, except in case of symptomatic HIV disease and/or an AIDS-defining illness.
* HIV-2 co infection.
* Use of co-medication with a known pharmacological interaction which precludes the appropriate use of one or more of the study drugs.
* Anticipated non-compliance with the protocol.
* Presence of a newly (within 30 days prior to the time of enrolment) diagnosed HIV-related opportunistic infection or condition which may interfere with the ability to comply with the study.
* Chronic active viral hepatitis or other chronic liver disease, which in the opinion of the investigator is a contraindication for the use of any of the study drugs. Patients who may be considered to have active HBV replication (HBV-surface antigen positive and/or HBV-DNA positive) may be excluded in case the investigator feels that the benefit of starting tenofovir/emtricitabine does not outweigh the risk of a "hepatitis flare" in case tenofovir/emtricitabine would need to be prematurely discontinued for any reason during the trial. Chronic hepatitis C is allowed, provided that treatment for hepatitis C is not anticipated during the study period.
* Women who are pregnant, or have the intention to become pregnant during the study period.
* Clinically relevant laboratory abnormalities: anaemia, thrombocytopenia, leucopenia, elevated liver transaminases, elevated bilirubin, elevated amylase, elevated lipase, which in the opinion of the investigator is a contraindication for the use of any of the study drugs, or any current known clinical or laboratory parameter of ACTG Grade 4 (see Appendix 2). However, asymptomatic Grade 4 abnormalities will be permitted at the discretion of the investigator if deemed clinically appropriate. Abnormalities deemed insignificant by the investigator must be discussed with the sponsor prior to enrolment.
* Significant renal dysfunction (creatinine clearance [CrCl] <60 mL/min) and/or hepatic impairment (aspartate aminotransferase/alanine aminotransferase [AST/ALT] >3 X ULN and/or documented liver cirrhosis)

Note: The site will calculate each patient's CrCl using the Cockcroft-Gault formula as shown below:

CrCl = [140 - age (yr)] × weight (kg) × constant 72 × serum creatinine (Cr) (mg/dL) where, constant = 1 for men and 0.85 for women.

* Use of nephrotoxic agents which in the opinion of the investigator are a contraindication for the use of tenofovir disoproxil fumarate and any other of the study drugs.
* Patients who have received within 4 weeks prior to entry, or who have an anticipated need for treatment with radiation therapy or cytotoxic chemotherapeutic agents during the protocol study period.
* Patients who have taken any investigational drug 30 days prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-07; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To assess the differences in changes in plasma lipids after once-daily saquinavir/ritonavir (2000/100 mg) or atazanavir/ritonavir (300/100 mg) each in combination with tenofovir disoproxil fumarate (300 mg QD) and emtricitabine (200 mg QD) for 24 weeks

SECONDARY OUTCOMES:
To assess the differences in changes in plasma lipids after once-daily saquinavir/ritonavir (2000/100 mg QD) or atazanavir/ritonavir (300/100 mg QD) each in combination with tenofovir disoproxil fumarate and emtricitabine for 48 weeks.
To compare differences in changes in glucose metabolism.
To compare changes in fat redistribution in both study arms.
To relate differences in changes in lipids, glucose metabolism and abdominal fat distribution to the plasma exposure of the different protease inhibitors (including ritonavir) used in the trial.
To assess the change in estimated glomerular filtration rate (GFR) by Cockcroft-Gault, MDRD and cystatin C-derived equations in both study arms.
To compare the antiviral efficacy of both regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reiss, MD, PhD, Study Chair — Academic Medical Centre, University of Amsterdam, the Netherlands
Locations (1):
- Academic Medical Centre, University of Amsterdam, Amsterdam, Netherlands